CLINICAL TRIAL: NCT03060174
Title: The Influence of Non-medication-based Prophylaxis of Postoperative Delirium on Postoperative Delirium and Cognitive Deficit
Brief Title: Study of Prevention of Postoperative Delirum to Reduce Incidence of Postoperative Cognitive Dysfunction
Acronym: DelPOCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PV4654
Record Dates: First submitted 2014-06-16; First posted 2017-02-23 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Delirium
MeSH Terms: conditions — Postoperative Cognitive Complications; Emergence Delirium

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- monitoring and non-medical prophylaxis of delirium (Other): The treatment group will receive monitoring and prophylaxis of delirium. The study arm designed to prevent delirium incorporates reorientation (watches, calendar, family photos, use of hearing aids, glasses and dentures, cognitive stimulation (newspaper, magazines, radio, television), early mobilisation, early enteral nutrition, early removal of drains or catheters, normalizing sleep-awake-rhythm.
  Interventions: Other: monitoring and non-medical prophylaxis of delirium
- Standard (No Intervention): The standard group will receive standard monitoring and standard treatment. The indication, choice and dosage of the medication used to treat delirium will be at the discretion of the ward doctor and will not be influenced by this study. The chosen medication as well as its dosage will be documented.

INTERVENTIONS:
Other: monitoring and non-medical prophylaxis of delirium
  Arms: monitoring and non-medical prophylaxis of delirium

SUMMARY:
Postoperative cognitive dysfunction describes a condition where cognitive functions such as attention, perception, concentration, learning, abstract thinking and problem solving are impaired postoperatively. These changes can be resolved after weeks and months, but in some cases may be permanent.

The aetiology is multifactorial. One risk factor for developing POCD is the occurrence of postoperative delirium.

A total of 638 consecutive patients will be enrolled in the study. Patients will be followed up at 7 days, 3 months and 1 year postoperatively. The cognitive function will be tested and compared to tests done before surgery. Postoperatively (from the day of operation until the 7th day and except of day 6) the grade of sedation; agitation; signs of delirium; pain; cardiac; respiratory; renal and infectious complications will be recorded.

As possible influencing factors, the investigators will document diagnosed depression; comorbidities; intraoperative blood loss; length of hospital stay; 1-year-mortality; number of operations/anaesthetics undergone after the initial operation.

Parameters that could trigger either depressive symptoms, neurocognitive dysfunction, anxiety, fatigue or lack of concentration will be recorded. These include: anaemia, hypercalcaemia, thyroidal gland hormones, electrolytes, creatinine, urea, glomerular filtration rate, cortisone therapy and adrenal cortical insufficiency.

DETAILED DESCRIPTION:
The methods include a neuropsychological test battery: TAP 2.3 (attention), Trail Making Test (TMT )A+B (attention), Digit span (memory), (Visual Learning and Memory Test (VLMT) (memory), Regensburgerwortfluessigkeitstest/fluency (RWT) subtests (executive function), Mehrfach-Wortschatz-Intelligenztest/vocabulary (MWT-B) (premorbid IQ).

Other measures are Hospital Anxiety and Depression Scale (HADS-D) (depressive symptoms and anxiety), Mini Mental State Examination (MMSE) 2 (dementia), Confusion Assessment Method (CAM-ICU) (delirium), Richmond Agitation and Sedation Scale (RASS) (sedation and agitation), Numeric Rating Scale (NRS) (pain) and Short Form Health Survey (SF-12) (health related quality of life).

ELIGIBILITY:
Inclusion Criteria:

* Age > 60 years
* Cardiac surgery (on-pump/off-pump, standard/minimal invasive)
* Written informed patient's consent

Exclusion Criteria:

* Non-German speaking or not their first language
* Illiteracy
* Mental disability
* Non-corrigible vision impairment
* Non-corrigible hearing impairment
* Illegal substance abuse (current or past history)
* Alcohol abuse (current or past history)
* Chronic benzodiazepine use
* Psychosis (current or past history)
* Parkinson Disease
* Dementia
* Multiple sclerosis
* Epilepsy (current or past history)
* Cerebral tumor (current or past history)
* Apoplexy or intracranial bleeding (current or past history)
* Severe traumatic brain injury (current or past history)
* Severe liver disease (Child Pugh B, C, liver insufficiency)
* Severe kidney disease with dialysis
* Mini Mental Status Examination < 24 points

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Estimated)
Dates: Start 2014-05; Primary Completion 2018-05 (Actual); Study Completion 2021-05 (Actual)

PRIMARY OUTCOMES:
postoperative cognitive deficit (POCD) | change from baseline in cognitive function at day 7, 3 months and 1 year after operation
  measured by neuropsychological test battery, analysis

SECONDARY OUTCOMES:
incidence and severity of postoperative delirium | from the day of operation until the 7th postoperative day
  measured 3 times per day via CAM-ICU
number of patients with cardiac complications | day of operation until 7th postoperative day
  daily documentation of cardiac complications (central venous oxygen saturation, myocardial infarction, acute heart failure, others)
length of hospital stay | from day of admission until day of discharge, up to 24 weeks
mortality | 1 year
health related quality of life | 3 months, 1 year after operation
  Short Form Health Survey (SF-12)
number of patients with respiratory complications | day of operation until 7th postoperative day
  daily documentation of pulmonary complications (pneumonia, pulmonary oedema, others),
number of patients with renal complications | day of operation until 7th postoperative day
  daily documentation of renal complications (creatinine, haemo(dia)filtration or haemodialysis)
number of patients with complications in the immunosystem | day of operation until 7th postoperative day
  daily documentation of parameters mirroring the immune answer (C-reactive protein, leukocytes, procalcitonin)

OTHER OUTCOMES:
anxiety and depressive symptoms on HADS-D | 7 days, 3 months, 1 year after operation
  The Hospital Anxiety and Depression Scale (HADS-D) is used to measure depressive symptoms. The 7 items are answered on a 4-point scale from 0 to 3 with a scale score varying between 0 and 21 (0-7 = normal, 8-10 = borderline, 11-14 = severe depressive symptoms, >15 very severe depressive symptoms).
postoperative pain scores on the numeric rating scale (NRS) | day of operation until 7th postoperative day, 3 months, 1 year after operation
  scale
haemoglobin (Anaemia) on a score | intraoperative
  Score Hb < 6 g/dl, 6-7.99 g/dl, 8-9.99 g/dl, > 9.99 g/dl
blood loss | intraoperative
  estimated blood loss in milliliter

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology and Intensive Care Medicine, University Hospital Hamburg Eppendorf, Univ.-Prof. Dr. med. Alwin E. Goetz and Prof. Dr. med. Christian Zoellner, Hamburg, Germany